CLINICAL TRIAL: NCT03260192
Title: Circulating Tumor DNA to Monitor Response to Neoadjuvant Chemotherapy in Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Liu Qiang, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: LQBC020
Record Dates: First submitted 2017-08-14; First posted 2017-08-24 (Actual); Last update posted 2024-01-10 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer
Keywords: circulating tumor DNA
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. plasma separated within 2 hours in EDTA tubes, stored in -80 celsius refrigerator;
  2. plasma in Streck tube, shipped within 3 days to the lab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigators aim to investigate whether circulating tumor DNA is a sensitive marker to evaluate patients' response to neoadjuvant chemotherapy

DETAILED DESCRIPTION:
Neoadjuvant chemotherapy(NAC) is traditionally for locally advanced disease, converting an inoperable to a resectable tumor.In recent years, it has become an option for patients of lower tumor stage to increase the possibility of breast conserving therapy. An effective method to monitor the response to NAC is important.

ELIGIBILITY:
Inclusion Criteria:

* Female patients undergoing NAC
* Age: 18-70 yrs
* Any menopausal status
* Any hormal receptor status

Exclusion Criteria:

* Metastasis discovered during NAC
* Lost more than 2 blood samples during NAC and surgery

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patient receiving NAC
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2013-09-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
death of breast cancer | Follow-up time is estimated to be up to 5 years. The duration is from the date of diagnosis to date of death of breast cancer or date of death of any cause, whichever come first.
  The event is defined as death of breast cancer, which is a separate measure

SECONDARY OUTCOMES:
tumor recurrence or distant metastasis | Follow-up time is estimated to be up to 5 years.The duration is from diagnosis to local recurrence or distant metastasis of breast cancer. Patients were followed up every six months in first three years, then followed up once a year.
  The event is defined as breast cancer local recurrence or distant metastasis

CONTACTS AND LOCATIONS:
Overall Officials: qiang Liu, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sunyat-sen Memorial Hospital, Guandong, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided